CLINICAL TRIAL: NCT03424330
Title: Evaluation of ReX-C System in Measurement and Improvement of Adherence, in Patients Receiving Oral Anti-coagulation Therapy for the Treatment and Prevention of Thromboembolism.
Brief Title: Evaluation of ReX-C System in Measurement and Improvement of Patients' Adherence.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dosentrx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RXC-154-2017-CLE
Record Dates: First submitted 2018-01-15; First posted 2018-02-07 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study will employ a randomized, controlled crossover study design.
  The study comprises two stages:
  * Stage 1: ReX-C Intervention in which subjects will use ReX-C to receive medication.
  * Stage 2: Control, in which Treatment as Usual (TAU). All subjects enrolled for the study will participate in both stages in a randomized crossover mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1 - ReX first (Experimental): Subjects begin with the ReX-C Intervention stage followed by Standard of Care stage.
  Interventions: Device: ReX-C intervention; Other: Standard of Care
- Arm 2- Standard of Care first (Experimental): Subjects start with Standard of Care stage followed by ReX-C Intervention.
  Interventions: Device: ReX-C intervention; Other: Standard of Care

INTERVENTIONS:
Device: ReX-C intervention — Patients receive medication by the ReX-C device
Other: Standard of Care — Patients receive medication as usual

SUMMARY:
The study aims to evaluate the safety, usability and efficacy of the ReX-C - a novel medication management system - in measurement and improvement of adherence, in patients receiving oral anti-coagulation therapy for the treatment and prevention of thromboembolism.

DETAILED DESCRIPTION:
ReX-C is a mobile system intended to provide solid, oral medication on patient demand, according to a pre-programmed treatment protocol. ReX-C addresses poor adherence to medication therapy by providing real-time, reliable adherence data to caregivers and timely, personalized reminders to patients.

During the study, the use of ReX-C system to receive medications will be compared to Standard of Care. Patients' adherence will be evaluated for both methods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, at least 18 years of age
2. Subject is able to swallow pills and use ReX-C device to receive medication.
3. Subject is able to read and understand the Informed Consent Form.
4. Subject receives anti-coagulants for the treatment and prevention of thromboembolism events, (e.g: Arterial Fibrillation (AF), Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)).
5. Subject receives Novel Oral Anti-coagulant (NOAC); including; Pradaxa® (dabigatran), Xarelto® (rivaroxaban) and Eliquis® (apixaban).

   1. Subject is recruited at least 1 month after treatment initiation and has stable dose regime.
   2. Subject receives stable dose of medication for at least a month.
6. Subject takes medication therapy at home.

Exclusion Criteria:

1. Subject has significant physical disability including; poor fine motor skills, impaired visual or auditory faculties, mental disorders or other impairment affecting ability to provide Informed Consent Form or use the ReX-C dispensing unit effectively.
2. Subject cen not use ReX-C to receive medications.
3. Subject is participating in another clinical study that does not permit participation in two studies simultaneously.
4. Subject is at end stage or terminal illness with anticipated life expectancy of 6 months or less.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Safety of ReX- C system, measured by incidences of pill overdose, pills malformation and adverse events related to the device use. | 18 weeks
  incidences of pill overdose, pills malformation and adverse events related to the device use will be measured by a questionnaire.
Ease of use and acceptance of ReX-C system measured by a questionnaire | 18 weeks
  Patients will be asked about their experience with ReX-C.
ReX-C capability to assess patient's adherence, measured by ReX-C record of missed/ delayed dose. | 18 weeks
  Any event of delayed pill intake recorded by ReX-C should lead to a personal reminder to patient, who has to confirm the delay and act to take the missing dose.

SECONDARY OUTCOMES:
Adherence rate measured by patient's plasma drug level | 18 weeks
  A comparison of adherence rate, measured by patient's plasma drug level, between ReX intervention stage and Standard of Care stage

CONTACTS AND LOCATIONS:
Overall Officials: Meir Preis, MD, Principal Investigator — Carmel Medical Center, Haifa, Israel
Locations (1):
- Carmel Medical Center, Haifa, Israel